CLINICAL TRIAL: NCT03774654
Title: Allogeneic Natural Killer T-Cells Expressing CD19 Specific Chimeric Antigen Receptor and Interleukin-15 in Relapsed or Refractory B-Cell Malignancies
Brief Title: CD19.CAR Allogeneic NKT for Patients With Relapsed or Refractory B-Cell Malignancies (ANCHOR)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Center for Cell and Gene Therapy, Baylor College of Medicine (Other); The Methodist Hospital Research Institute (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Carlos Ramos, Associate Professor, Baylor College of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-44526 ANCHOR; P50CA126752 (NIH)
Record Dates: First submitted 2018-12-11; First posted 2018-12-13 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Refractory B-Cell Non-Hodgkin Lymphoma; Refractory B-Cell Small Lymphocytic Lymphoma; Relapsed Adult ALL; Relapsed CLL; Relapsed Non Hodgkin Lymphoma
Keywords: Gene Therapy; CAR T-cells; chimeric antigen receptor; B-Cell Malignancies; CD19
MeSH Terms: conditions — Lymphoma, B-Cell; Leukemia, B-Cell; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- CD19.CAR-aNKT cells (cohort A, non-ALL) (Experimental): This cohort is for patients without refractory/relapsed B-cell NHL or leukemia (ALL). Three dose levels will be evaluated. Patients will also receive lymphodepletion chemotherapy consisting of cyclophosphamide and fludarabine followed by the CD19.CAR-aNKT cell infusion.
  Interventions: Genetic: CD19.CAR-aNKT cells
- CD19.CAR-aNKT cells (cohort B, ALL). (Experimental): This cohort is for patients with refractory/relapsed B-cell NHL or leukemia (ALL). Three dose levels will be evaluated. Patients will also receive lymphodepletion chemotherapy consisting of cyclophosphamide and fludarabine followed by the CD19.CAR-aNKT cell infusion.
  Interventions: Genetic: CD19.CAR-aNKT cells

INTERVENTIONS:
Genetic: CD19.CAR-aNKT cells — Patients will be given the T-cell product by intravenous injection (into the vein through an IV line) at the assigned dose..
  Dose Level 1: 1 x 10^7/m2. Dose Level 2: 3 x 10^7/m2. Dose Level 3: 1 x 10^8/m2. Dose Level 4: 3 x 10^8/m2.

SUMMARY:
This study is for patients who have lymphoma or leukemia that has come back or has not gone away after treatment. Because there is no standard treatment for this cancer, patients are being asked to volunteer for a gene transfer research study using special immune cells.

The body has different ways of fighting infection and disease. No single way seems perfect for fighting cancers. This research study combines two different ways of fighting disease, antibodies and immune cells. Antibodies are types of proteins that protect the body from bacteria and other diseases. Immune cells, also called lymphocytes, are special infection-fighting blood cells that can kill other cells including tumor cells. Both antibodies and lymphocytes have been used to treat patients with cancer. They have shown promise, but have not been strong enough to cure most patients.

The antibody used in this study is called anti-CD19. This antibody sticks to lymphoma cells because of a substance on the outside of the cells called CD19. CD19 antibodies have been used to treat people with lymphoma and leukemia. For this study, the anti-CD19 antibody has been changed so that instead of floating free in the blood it is now joined to the NKT cells, a special type of lymphocytes that can kill tumor cells but not very effectively on their own. When an antibody is joined to a T cell in this way it is called a chimeric receptor. Investigators have also found that NKT cells work better if proteins are added that stimulate lymphocytes, such as one called CD28. Adding the CD28 makes the cells last for a longer time in the body but maybe not long enough for them to be able to kill the lymphoma cells. It is believed that by adding an extra stimulating protein, called IL-15, the cells will have an even better chance of killing the lymphoma cells.

In this study the investigators are going to see if this is true by putting the anti-CD19 chimeric receptor with CD28 and the IL-15 into NKT cells grown from a healthy individual. These cells are called ANCHOR cells. These cells will be infused into patients that have lymphomas or leukemias that have CD19 on their surface. The ANCHOR cells are investigational products not approved by the Food and Drug Administration.

The purpose of this study is to find the biggest dose of ANCHOR cells that is safe, to see how long the ANCHOR cells last, to learn what their side effects are and to see whether this therapy might help people with lymphoma or leukemia.

DETAILED DESCRIPTION:
Earlier, a healthy donor provided blood to make ANCHOR cells in the laboratory. These cells were grown and frozen for later use. To make the ANCHOR cells, the investigators took the donor blood and stimulated it with growth factors to make the NKT cells grow. To get the CD19 antibody, CD28 and IL-15 into the NKT cells, they were infected with a virus, called a retrovirus. This virus cannot grow and infect other cells, but delivered a new genetic message into the ANCHOR cells that provides the instructions for the cells to make the CD19 antibody, CD28 and IL-15. This new genetic message will also help the investigators to find the ANCHOR cells in the blood after they are injected. Because patients will have received cells with a new gene in them, patients will be followed for a total of 15 years to see if there are any long term side effects of gene transfer.

Patients will be assigned a dose of ANCHOR cells. This is a dose escalation study. This means that at the beginning, patients will be started on the lowest dose of ANCHOR cells. Once that dose schedule proves safe, the next group of patients will be started at a higher dose. This process will continue until all 4 dose levels are studied. If the side effects are too severe, the dose will be lowered or the infusions will be stopped.

In this study, patients will receive treatment with cyclophosphamide and fludarabine. These drugs will decrease the numbers of the patients own immune cells before the ANCHOR cells are infused.

The patient will be given an injection of ANCHOR cells into the vein through an IV at the assigned dose. Before receiving the injection, the patient may be given a dose of Benadryl and Tylenol. The injection will take about 20 minutes. The patient will then be monitored in the clinic for up to 2 hours. Certain patients with aggressive lymphomas will need to be admitted to the hospital for the first three days after receiving the cells. Patients will need to stay in Houston for 4 weeks after the ANCHOR cell infusion to monitor them for side effects. Patients will have follow-up visits 3 times per week at weeks 1, 2, 3, 4, and once during week 6; months 3, 6, 9, and 12; twice a year for 4 years and then once a year for the next 10 years - for a total of 15 years). Patients will also have scheduled disease evaluations after the ANCHOR cell infusion (at week 4 and then as clinically needed).

The treatment will be given by the Center for Cell and Gene Therapy in Texas Chidren's Hospital or Houston Methodist Hospital.

Medical tests before treatment--

Before being treated, the patient will receive a series of standard medical tests:

* Physical exam and History
* Blood tests to measure blood cells, kidney and liver function
* Measurements of tumor by scans and/or bone marrow studies
* A urine or serum pregnancy test, when applicable

Medical tests during and after treatment--

Patients will receive standard medical tests when getting the infusions and afterwards. The evaluations that will be done at these visits include:

* Physical exams and History
* Blood tests to measure blood cells, kidney and liver function
* Measurements of the tumor by scans at 4-6 weeks, 3 months, 6 months, 9 months and 12 months
* If you have disease in the bone marrow, measurements of your tumor by bone marrow studies at 8-12 weeks, 6 months, 9 months and 12 months after the infusion.
* To learn more about the way the ANCHOR cells are working and how long they last in the body, extra blood will be drawn. On the day patients receive the cells, blood will be taken before the cells are given and a few hours afterwards. Other blood will be drawn one week after the infusion, 2 weeks, 3 weeks (optional), 4 weeks, and 6 weeks after the infusion, at 3 months, at 6 months, at 9 months, at 1 year, twice a year for 4 years, then yearly for the next 10 years - for a total of 15 years.

During the time points listed above, if the ANCHOR cells are found in the patient's blood above a certain amount, an extra 5 mL of blood may need to be collected for additional testing.

If the patient has a biopsy of a lymph node, like a repeat tumor or bone marrow study, the investigators may ask to have a piece for research purposes.

Patients will receive supportive care for any acute or chronic toxicities, including blood components or antibiotics, and other intervention as appropriate.

ELIGIBILITY:
Treatment Inclusion Criteria:

1. Diagnosis of CD19-positive B-cell lymphoma or leukemia (ALL or CLL).
2. The disease is:

   Cohort A (non-ALL patients):
   1. Relapsed or refractory after two or more lines of therapy, including a CD20 antibody, if an indolent lymphoma.
   2. Relapsed or refractory after two or more lines of therapy, including ibrutinib and venetoclax, if CLL.
   3. Relapsed or refractory after two or more lines of therapy, including a CD20 antibody and an anthracycline, and the patient is ineligible for autologous stem cell transplantation, if an aggressive or highly aggressive lymphoma.

      * Ineligibility for autologous stem cell transplantation includes non-responsive disease after salvage therapy and failure to mobilize stem cells for transplant.

   Cohort B (ALL patients)

   a. Relapsed or refractory after two or more lines of therapy, if ALL.
3. Measurable disease by current criteria (Lugano criteria for lymphomas, IWG criteria for CLL, and detectable disease for ALL).
4. Age ≥ 3 and ≤75 years.
5. Bilirubin < 2 times (3 times if Gilbert syndrome) upper limit of normal
6. AST and ALT less than 5 times the upper limit of normal.
7. Estimated GFR ≥ 50 mL/min.
8. Pulse oximetry of ≥ 90% on room air
9. Karnofsky or Lansky score of ≥ 70.
10. Recovered from the acute toxic effects of all prior chemotherapy based on the enrolling physician's assessment (if some effects of chemotherapy are expected to last long term, patient is eligible if meeting other eligibility criteria).
11. Life expectancy of greater than 12 weeks.
12. Sexually active patients must be willing to utilize one of the more effective birth control methods during the study and for 6 months after the study is concluded. The male partner should use a condom.
13. Patients must sign an informed consent indicating that they are aware this is a research study and have been told of its possible benefits and toxic side effects. Patients or their guardians will be given a copy of the consent form.

Treatment Exclusion Criteria:

1. Currently receiving any investigational agents or received any cellular therapies within the previous 6 weeks.
2. History of hypersensitivity reactions to murine protein-containing products.
3. History of grade 2 to 4 graft-versus-host disease (GVHD)
4. Pregnant or lactating.
5. Active infection with HIV or HTLV.
6. Active infection with HBV or HCV.
7. Uncontrolled active bacterial, fungal or other viral infection.

Ages: 3 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2020-06-22 (Actual); Primary Completion 2026-06-20 (Estimated); Study Completion 2035-02-28 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) rate | 4 weeks post T cell infusion
  DLT rate is defined as the proportion of subjects with DLT evaluated as per the NCI CTCAE v5.0 with the exception of CRS and neurological toxicities that are related to T-cell infusions. GVHD will be graded according to the BMT CTN Technical Manual of Procedures v3.0.

SECONDARY OUTCOMES:
Frequency of circulating CD19.CAR-aNKT cells transduced with the vector. | 6 weeks post T cell infusion
  The frequency of the infused cells will be summarized at pre- and post-infusion time points to evaluate their expansion and persistence.
Overall response rate according to the Lugano criteria for non-Hodgkin lymphomas (for NHL) and the IWG (for CLL), or the proportion of patients with morphologic CR (for ALL). | 4-6 weeks post T cell infusion
  Overall response rate is defined as the proportion of subjects with best overall response of complete response (CR) or partial response (PR) according to the Lugano criteria for non-Hodgkin lymphomas (for NHL) and the IWG (for CLL), or the proportion of patients with morphologic CR (for ALL).

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Ramos, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Houston Methodist Hospital, Houston, Texas
  - Texas Children's Hospital, Houston, Texas